CLINICAL TRIAL: NCT00643682
Title: Improving Bowel Preparation for Colonoscopy With a Simple Educational Card
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Brian Jacobson, Associate Professor of Medicine, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BMC-GI-1
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Results first posted 2012-10-01 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-08

CONDITIONS: Colonic Polyps; Colonic Neoplasms
Keywords: colonoscopy; bowel preparation; patient education; polyp detection
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Patients in this arm will be given an educational card in addition to the standard pre-endoscopy instructions.
  Interventions: Other: Educational card
- B (No Intervention): Patients in this arm will be given the standard pre-endoscopy instructions.

INTERVENTIONS:
Other: Educational card — A 4x6 inch educational card containing a photo of an unprepared colon and a clean colon with the caption: "Drinking all the bowel cleaning medicine as described in the enclosed instructions lets the doctor see your colon better during your colonoscopy."
  Arms: A

SUMMARY:
The purpose of this study is to determine whether adding a simple educational card to standard pre-procedure instructions improves the quality of bowel preparation for colonoscopy.

DETAILED DESCRIPTION:
Despite written instructions, many patients do not understand the importance of bowel preparation as they prepare for colonoscopy. This often leads to poor compliance with preparation protocol and therefore inadequate bowel preparation. Our goal is to include a simple educational card which will hopefully improve the quality of bowel preparation by providing a visual component with the preparation instructions. This card will stress the importance of drinking the entire bowel preparation and provide representative images of a dirty and clean colon. We will specifically target patients directly booked for screening colonoscopy (those without a pre-procedure office visit). In a randomized fashion, patients in the control group will receive the standard bowel preparation instructions and patients in the intervention group will receive the educational card along with the standard bowel preparation instructions. The primary outcome will be the endoscopist's assessment of the quality of preparation using a standardized bowel preparation scale. Secondary outcomes will include the number and types of polyps found, colonoscope insertion and withdrawal time, and patient satisfaction with the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* 18 years old or older
* Referred and scheduled for an elective screening colonoscopy

Exclusion Criteria:

* Inpatients
* Prisoners
* Cognitively impaired patients
* Legally blind patients
* Patients allergic to polyethylene glycol electrolyte lavage solution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2006-02; Primary Completion 2008-06 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian C Jacobson, MD, MPH, Principal Investigator — Boston University
Locations (1):
- Boston University Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Calderwood AH, Lai EJ, Fix OK, Jacobson BC. An endoscopist-blinded, randomized, controlled trial of a simple visual aid to improve bowel preparation for screening colonoscopy. Gastrointest Endosc. 2011 Feb;73(2):307-14. doi: 10.1016/j.gie.2010.10.013. Epub 2010 Dec 18. PMID 21168840

RESULTS

PARTICIPANT FLOW:
Groups:
- Educational Card: Patients in this arm will be given an educational card in addition to the standard pre-endoscopy instructions.
- Control: Patients in this arm will be given the standard pre-endoscopy instructions.
Period: Overall Study
Arm/Group | Educational Card | Control
Started | 999 | 1001
Completed | 477 | 492
Not Completed | 522 | 509
Not completed — did not keep appointment | 522 | 509

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Educational Card | Control | Total
Number analyzed (Participants) | 477 | 492 | 969
Age Continuous [Mean (Standard Deviation); unit: years] | 57 (8) | 57 (7) | 57 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 279 | 287 | 566
  Male | 198 | 205 | 403
Region of Enrollment [Number; unit: participants]
  United States | 477 | 492 | 969

OUTCOME MEASURES:

1. Primary Outcome: Boston Bowel Preparation Scale Score
Description: An ordinal scale. 0=fully unprepared colon and 9=perfectly clean colon. Higher values represent a better outcome. For reference please see: Lai EJ, Calderwood AH, Doros G, Fix OK, Jacobson BC. The Boston bowel preparation scale: a valid and reliable instrument for colonoscopy-oriented research. Gastrointestinal Endoscopy 2009;69:620-625. PMCID: PMC2763922
Time Frame: 2 years
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Educational Card | Control
Number analyzed (Participants) | 477 | 492
units on a scale | 6 [6 to 7] | 6 [6 to 7]

2. Secondary Outcome: Time to Advance Colonoscope From Anus to Tip of Cecum.
Description: time in minutes to advance colonoscope from anus to tip of cecum during insertion phase of colonoscopy.
Time Frame: 2 years
Measure: Median (Inter-Quartile Range); unit: time in minutes
Arm/Group | Educational Card | Control
Number analyzed (Participants) | 477 | 492
time in minutes | 7 [5 to 10] | 7 [5 to 10]

3. Secondary Outcome: Time to Withdraw Colonoscope From Tip of Cecum to Anus.
Description: Time in minutes to withdraw colonoscope from tip of cecum to anus during withdrawal phase of colonoscopy
Time Frame: 2 years
Measure: Median (Inter-Quartile Range); unit: Time in minutes
Arm/Group | Educational Card | Control
Number analyzed (Participants) | 477 | 492
Time in minutes | 8 [6 to 11] | 7 [6 to 10]

4. Secondary Outcome: Number of Repeat Procedures Recommended Due to Inadequate Bowel Preparation.
Description: The number of times a colonoscopist recommended that the bowel was too unclean to qualify as an acceptable colonoscopy and therefore recommended repeating the procedure after better cleansing. This is both the number of participants with an inadequate preparation and the number of inadequate procedures. These are synonymous.
Time Frame: 2 years
Measure: Number; unit: participants who had a colonoscopy
Arm/Group | Educational Card | Control
Number analyzed (Participants) | 477 | 492
participants who had a colonoscopy | 51 | 49

ADVERSE EVENTS:
Arm/Group | Educational Card | Control
Serious Adverse Events (participants affected / at risk) | 0/477 | 0/492
Other Adverse Events (participants affected / at risk) | 0/477 | 0/942

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes